CLINICAL TRIAL: NCT03180762
Title: A 3-Part, Randomized, Placebo-controlled, Double-blind, Single Ascending Dose Study to Investigate Safety and Tolerability, Pharmacokinetics and Pharmacodynamics of JNJ-64140284 in Healthy Subjects
Brief Title: A Study to Investigate Safety and Tolerability, Pharmacokinetics and Pharmacodynamics of JNJ-64140284 in Healthy Participants
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Trial stopped: A SAE has occured. As a measure of precaution, the trial has been stopped.
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: CR108318; 2017-000283-16 (EudraCT Number); 64140284EDI1001 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2017-05-30; First posted 2017-06-08 (Actual); Last update posted 2018-10-30 (Actual); Status verified 2018-10

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Part 1: Cohort 1 (JNJ-64140284 or Placebo) (Experimental): Participants will receive 0.1 milligram (mg) JNJ-64140284 or matching placebo under fasted condition on Day 1.
  Interventions: Drug: JNJ-64140284 0.1 mg; Drug: Placebo
- Part 1: Cohort 2 (JNJ-64140284 or Placebo) (Experimental): Participants will receive 0.5 mg JNJ-64140284 or matching placebo under fasted condition on Day 1.
  Interventions: Drug: JNJ-64140284 0.5 mg; Drug: Placebo
- Part 1: Cohort 3 (JNJ-64140284 or Placebo) (Experimental): Participants will receive 2.5 mg JNJ-64140284 or matching placebo under fasted condition on Day 1.
  Interventions: Drug: JNJ-64140284 2.5 mg; Drug: Placebo
- Part 1: Cohort 4 (JNJ-64140284 or Placebo) (Experimental): Participants will receive 10 mg JNJ-64140284 or matching placebo under fasted condition on Day 1.
  Interventions: Drug: JNJ-64140284 10 mg; Drug: Placebo
- Part 1: Cohort 5 (JNJ-64140284 or Placebo) (Experimental): Participants will receive 50 mg JNJ-64140284 or matching placebo under fasted condition on Day 1.
  Interventions: Drug: JNJ-64140284 50 mg; Drug: Placebo
- Part 1: Cohort 6 (JNJ-64140284 or Placebo) (Experimental): Participants will receive 150 mg JNJ-64140284 or matching placebo under fasted condition on Day 1.
  Interventions: Drug: JNJ-64140284 150 mg; Drug: Placebo
- Part 2: Cohort 7 (JNJ-64140284) (Experimental): Participants will receive JNJ-64140284 (dose to be determined - the dose of JNJ-64140284 will be determined on the basis of acceptable safety, tolerability and pharmacokinetics [PK] of preceding dose levels; no more than 50 percent (%) of the highest dose tested [though as high as possible within this restriction] and considered well tolerated in Part 1) under fed conditions on Day 1.
  Interventions: Drug: JNJ-64140284 (dose to be determined [TBD])
- Part 3: Cohort 8 (JNJ-64140284 or Placebo) (Experimental): Participants will receive JNJ-64140284 or matching placebo (dose to be determined - dose will be determined based on PK data from previous cohorts and which will be well-tolerated in Part 1) under fasted condition on Day 1.
  Interventions: Drug: JNJ-64140284 (dose to be determined [TBD]); Drug: Placebo

INTERVENTIONS:
Drug: JNJ-64140284 0.1 mg — 0.1 mg of JNJ-64140284 will be administered as an oral solution.
  Arms: Part 1: Cohort 1 (JNJ-64140284 or Placebo)
Drug: JNJ-64140284 0.5 mg — 0.5 mg of JNJ-64140284 will be administered as an oral solution.
  Arms: Part 1: Cohort 2 (JNJ-64140284 or Placebo)
Drug: JNJ-64140284 2.5 mg — 2.5 mg of JNJ-64140284 will be administered as an oral solution.
  Arms: Part 1: Cohort 3 (JNJ-64140284 or Placebo)
Drug: JNJ-64140284 10 mg — 10 mg of JNJ-64140284 will be administered as an oral solution.
  Arms: Part 1: Cohort 4 (JNJ-64140284 or Placebo)
Drug: JNJ-64140284 50 mg — 50 mg of JNJ-64140284 will be administered as an oral solution.
  Arms: Part 1: Cohort 5 (JNJ-64140284 or Placebo)
Drug: JNJ-64140284 150 mg — 150 mg of JNJ-64140284 will be administered as an oral solution.
  Arms: Part 1: Cohort 6 (JNJ-64140284 or Placebo)
Drug: JNJ-64140284 (dose to be determined [TBD]) — JNJ-64140284 (dose to be determined) will be administered as an oral solution.
  Arms: Part 2: Cohort 7 (JNJ-64140284); Part 3: Cohort 8 (JNJ-64140284 or Placebo)
Drug: Placebo — Matching placebo will be administered.
  Arms: Part 1: Cohort 1 (JNJ-64140284 or Placebo); Part 1: Cohort 2 (JNJ-64140284 or Placebo); Part 1: Cohort 3 (JNJ-64140284 or Placebo); Part 1: Cohort 4 (JNJ-64140284 or Placebo); Part 1: Cohort 5 (JNJ-64140284 or Placebo); Part 1: Cohort 6 (JNJ-64140284 or Placebo); Part 3: Cohort 8 (JNJ-64140284 or Placebo)

SUMMARY:
The purpose of this study is to investigate the safety and tolerability of JNJ-64140284 versus placebo after single oral dose administration (ascending dose levels) under fasted condition, to characterize the pharmacokinetics (PK) of JNJ-64140284 in plasma, cerebrospinal fluid (CSF) and urine after single oral dose administration and to investigate the effect of food (high fat/high calorie) on the PK of JNJ-64140284 following single oral dose administration.

ELIGIBILITY:
Inclusion Criteria:

Part 1 and 2:

- Healthy male participants between 18 and 58 years of age, inclusive

Part 1, 2 and 3:

- Participants must be healthy on the basis of clinical laboratory tests performed at screening. If the results of the serum chemistry panel, hematology, or urinalysis are outside the normal reference ranges, retesting of an abnormal lab value(s) that may lead to exclusion will be allowed once during the screening phase. The participant may be included only if the investigator judges the abnormalities or deviations from normal to be not clinically significant or to be appropriate and reasonable for the population under study according to both the investigator and to the Janssen Safety Physician, are acceptable

Part 3:

* Healthy male and female participants between 59 and 75 years of age, inclusive
* Participants must be healthy and medically stable on the basis of clinical laboratory tests (at screening) and physical and neurological examination (at screening and at admission to the clinical unit). If the participant is medically stable with medication, inclusion can be allowed on a case by case basis with written agreement of the sponsor's responsible safety physician
* Women must not be of childbearing potential (must be postmenopausal with amenorrhea for at least 12 months) or permanently sterilized (for example, tubal occlusion, hysterectomy, bilateral salpingectomy)

Exclusion Criteria:

Part 1, 2 and 3:

* Participants with a history of or current significant medical illness including (but not limited to) cardiac arrhythmias or other cardiac disease, hematological disease, lipid abnormalities, bronchospastic respiratory disease, diabetes mellitus, renal or hepatic insufficiency, thyroid disease, Parkinson's disease, infection, or any other illness that the Investigator considers should exclude the participant
* Participants with a serology positive for hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibodies or human immunodeficiency virus (HIV) antibodies
* Participants with a clinically significant acute illness within 7 days prior to study drug administration
* Donation of 1 or more units (approximately 450 milliliter [mL]) of blood or acute loss of an equivalent amount of blood within 90 days prior to study drug administration

Part 3:

- participants having a contraindication for spinal puncture including:

1. A relevant history of lower back pain or scoliosis or kyphosis and/or major (lumbar) back surgery (microdiscectomy is allowed) in the opinion of the investigator
2. Allergy to local anesthetics and/or iodine/disinfectants
3. Clinically significant abnormal values for coagulation at screening
4. Use of aspirin (even low dose) within 5 days prior to lumbar puncture
5. Use of low molecular weight heparin (LMWH) within 12 hours prior to lumbar puncture
6. Use of any anticoagulant treatment (besides LMWH described above) within 1 week prior to lumbar puncture
7. Has a topical infection or local dermatological condition at the puncture site prior to puncture
8. Has papilloedema or signs of increased intracranial pressure based on fundoscopy at screening

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2017-05-30 (Actual); Primary Completion 2017-09-25 (Actual); Study Completion 2017-09-25 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Adverse Events (AEs) as a Measure of Safety and Tolerability: Part 1, Part 2, and Part 3 | Approximately 40 days
  An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study.
Maximum Plasma Concentration (Cmax) of JNJ-64140284: Part 1, Part 2, and Part 3 | Predose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, 24, 36, 48, 72 and 96 hours post dose
  The Cmax is the maximum observed plasma concentration.
Maximum Cerebrospinal Fluid (CSF) Concentration (Cmax) of JNJ-64140284: Part 3 | Predose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, and 12 hours post dose
  The Cmax is the maximum observed CSF concentration.
Last Quantifiable Plasma Concentration (Clast) of JNJ-64140284: Part 1, Part 2, and Part 3 | Predose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, 24, 36, 48, 72 and 96 hours post dose
  The Clast is the last quantifiable plasma concentration.
Last Quantifiable CSF Concentration (Clast) of JNJ-64140284: Part 3 | Predose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, and 12 hours post dose
  The Clast is the last quantifiable CSF concentration.
Time to Reach Maximum Plasma Concentration (Tmax) of JNJ-64140284: Part 1, Part 2, and Part 3 | Predose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, 24, 36, 48, 72 and 96 hours post dose
  The Tmax is defined as actual sampling time to reach maximum observed plasma concentration.
Time to Reach Maximum CSF Concentration (Tmax) of JNJ-64140284: Part 1, Part 2, and Part 3 | Predose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, and 12 hours post dose
  The Tmax is defined as actual sampling time to reach maximum observed CSF concentration.
Time of the Last Quantifiable Plasma Concentration (Tlast) of JNJ-64140284: Part 1, Part 2, and Part 3 | Predose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, 24, 36, 48, 72 and 96 hours post dose
  The Tlast is defined as the time of the last quantifiable plasma concentration.
Time of the Last Quantifiable CSF Concentration (Tlast) of JNJ-64140284: Part 3 | Predose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, and 12 hours post dose
  The Tlast is defined as the time of the last quantifiable CSF concentration.
Area Under the Plasma Concentration-Time Curve From Time Zero to Time of the Last Quantifiable Concentration (AUC [0-last]) of JNJ-64140284: Part 1, Part 2, and Part 3 | Predose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, 24, 36, 48, 72 and 96 hours post dose
  The (AUC [0-last]) is the area under the plasma concentration-time curve from time 0 to time of the last quantifiable concentration.
Area Under the CSF Concentration-Time Curve From Time Zero to Time of the Last Quantifiable Concentration (AUC [0-last]) of JNJ-64140284: Part 1, Part 2, and Part 3 | Predose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, and 12 hours post dose
  The (AUC [0-last]) is the area under the CSF concentration-time curve from time 0 to time of the last quantifiable concentration.
Area Under the Plasma Concentration-Time Curve From Time Zero to Infinite Time (AUC [0-infinity]) of JNJ-64140284: Part 1, Part 2, and Part 3 | Predose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, 24, 36, 48, 72 and 96 hours post dose
  The AUC (0-infinity) is the area under the plasma concentration-time curve from time zero to infinite time, calculated as the sum of AUC(0-last) and C(0-last)/lambda(z), wherein AUC(0-last) is the area under the plasma concentration-time curve from time 0 to time of the last quantifiable concentrations; C(0-last) is the last observed quantifiable concentration; and lambda(z) is elimination rate constant.
Area Under the CSF Concentration-Time Curve From Time Zero to Infinite Time (AUC [0-infinity]) of JNJ-64140284: Part 3 | Predose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, and 12 hours post dose
  The AUC (0-infinity) is the area under the CSF concentration-time curve from time zero to infinite time, calculated as the sum of AUC(0-last) and C(0-last)/lambda(z), wherein AUC(0-last) is the area under the CSF concentration-time curve from time 0 to time of the last quantifiable concentrations; C(0-last) is the last observed quantifiable concentration; and lambda(z) is elimination rate constant.
Elimination Rate Constant (Lambda[z]) of JNJ-64140284: Part 1, Part 2, and Part 3 | Predose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, 24, 36, 48, 72 and 96 hours post dose
  Lambda(z) is first-order rate constant associated with the terminal portion of the curve, determined as the negative slope of the terminal log-linear phase of the drug concentration-time curve.
Elimination Half-life (t1/2) of JNJ-64140284: Part 1, Part 2, and Part 3 | Predose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, 24, 36, 48, 72, and 96 hours post dose
  The t1/2 is the time measured for the plasma concentration to decrease by 1 half to its original concentration. It is associated with the terminal slope of the semi logarithmic drug concentration-time curve, and is calculated as 0.693/lambda(z).
Total Clearance (CL/F) of JNJ-64140284: Part 1, Part 2, and Part 3 | Predose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, 24, 36, 48, 72 and 96 hours post dose
  CL/F is the total clearance of drug after extravascular administration, uncorrected for absolute bioavailability.
Creatinine Clearance (CLcr) of JNJ-64140284: Part 1, Part 2, and Part 3 | Predose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, 24, 36, 48, 72 and 96 hours post dose
  CLcr will be determined with the Cockcroft-Gault formula.
Amount of Drug Excreted in Urine From Time Zero to Infinite Time (Aeinf): Part 1 | 0-1, 1-2, 2-4, 4-12, and 12-24 hours post dose
  Aeinf is the cumulative amount of study drug excreted into urine from time of dosing extrapolated to time infinity.
Renal Clearance (CLr): Part 1 | 0-1, 1-2, 2-4, 4-12, and 12-24 hours post dose
  The CLr is the renal clearance of the drug.

SECONDARY OUTCOMES:
Bond & Lader Visual Analogue Scale (VAS) Score: Part 1 and Part 3 | Days -1, 1, 2 and 3
  The VAS is a participant rated scale, made up of 16 (items) pairs of alternative descriptors of mood and attention at either end of a 10 cm line. The item score ranges from 0 to 100, with a high score reflecting a high level of anxiety, sedation or dysphoria.
Karolinska Sleepiness Scale (KSS) Score: Part 1 and Part 3 | Days -1, 1, 2 and 3
  The KSS is a participant-reported assessment used to rate sleepiness on a scale of 1 to 9, ranging from 'extremely alert' (1) to 'very sleepy, great effort to keep awake, fighting sleep' (9).
Profile of Mood States (POMS) Score: Part 1 and Part 3 | Days -1, 1, 2 and 3
  The POMS is a self-administered scale that assesses individuals' mood states. This is a validated scale to measure positive and negative mood states. The POMS contains 30 items describing the feeling/mood state rated by participants on a 5-point scale (where, 0=not at all and 4=extremely). The greater the score, the greater the corresponding mood state.
Body Sway: Part 1 | Days -1, 1, 2 and 3
  Body sway will be used to measure body movements, providing a measure of postural stability. The method has been used to demonstrate effects of sleep deprivation, alcohol, and benzodiazepines. It will be measured either using a stabilometric platform or a pot string meter based on the Wright ataxiameter.
Cognitive Test Battery: International Shopping List Test (ISLT): Part 1 | Days -21 to -2, Day -1, and Day 1 (6 hours post dose)
  The ISLT is a measure of Verbal Learning. The test measures total number of correct responses remembering the word list on 3 consecutive trials at a single assessment. Higher score indicates better performance.
Cognitive Test Battery: Groton Maze Learning Test (GMLT): Part 1 | Days -21 to -2, Day -1, Day 1 (2, 4, 6, and 12 hours post dose), and Day 2 (24 hours post dose)
  GMLT is a measure of Executive Function and Spatial Learning. The test measures total number of errors made while locating and learning 28 step pathway hidden beneath a 10*10 grid on 5 consecutive trials during a single session. Lower score indicates better performance.
Cognitive Test Battery: Detection Task (DET): Part 1 | Days -21 to -2, Day -1, Day 1 (2, 4, 6, and 12 hours post dose), and Day 2 (24 hours post dose)
  DET is a measure of Psychomotor Function. The test measures speed of performance; mean of the log10 transformed reaction times for correct responses. Lower score indicates better performance.
Cognitive Test Battery: Identification Task (IDN): Part 1 | Days -21 to -2, Day -1, Day 1 (2, 4, 6, and 12 hours post dose), and Day 2 (24 hours post dose)
  IDN is a measure of Attention. The test measures speed of performance; mean of the log10 transformed reaction times for correct responses. Lower score indicates better performance.
Cognitive Test Battery: One Card Learning Task (OCL): Part 1 | Days -21 to -2, Day -1, Day 1 (2, 4, 6, and 12 hours post dose), and Day 2 (24 hours post dose)
  OCL is a measure of Visual Learning. The test measures accuracy of performance; arcsine transformation of the square root of the proportion of correct responses. Higher score indicates better performance.
Cognitive Test Battery: One Back Task (ONB): Part 1 | Days -21 to -2, Day -1, Day 1 (2, 4, 6, and 12 hours post dose), and Day 2 (24 hours post dose)
  ONB is a measure of Working Memory. The test measures speed of performance; mean of the log10 transformed reaction times for correct responses. Lower score indicates better performance.
Cognitive Test Battery: Groton Maze Learning Test (GMLT) Delayed Recall: Part 1 | Days -21 to -2, Day -1, and Day 1 (6 hours post dose)
  GMLT delayed recall is a measure of Delayed Spatial Memory. The test measures number of errors made while locating 28 step pathway hidden beneath a 10*10 grid after a delay. Lower score indicates better performance.
Cognitive Test Battery: International Shopping List Test Delayed (ISLT-D): Part 1 | Days -21 to -2, Day -1, Predose, Day 1 (6 hours post dose), and Day 2 (24 hours post dose)
  ISLT-D is a measure of Delayed Verbal Memory. The test measures total number of correct responses recalling the word list learned initially. Higher score indicates better performance.
Sheehan Irritability Scale (SIS) Score: Part 1 and Part 3 | Day -1, Day 1 (6 and 12 hours post dose), and Day 2 (24 hours post dose)
  The SIS is a 7-item self-report rating scale that assess symptoms of irritability, frustration, edginess/impatience, moodiness, anger with self, anger with others and temper during the past hour. Each item is assessed on an 11-point numeric rating scale ranging from 0 (not at all) to 10 (extremely). The SIS total score is calculated by summing of the scores for each of the 7 individual items and ranges from 0 to 70. A higher score indicates greater symptomatology.
Cerebrospinal Fluid (CSF) Biomarkers Level: Brain Derived Neurotrophic Factor (BDNF): Part 3 | Predose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12 hours post dose
  BDNF level in the CSF (a CSF biomarker) will be analyzed to evaluate the pharmacodynamic effect of JNJ-64140284.
Cerebrospinal Fluid (CSF) Biomarkers Level: Monoaminergic Neurotransmitters and Their Metabolites: Part 3 | Predose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12 hours post dose
  Monoaminergic neurotransmitters (such as dopamine, serotonine and [nor]adrenaline) and their metabolites (such as homovanillic acid [HVA], 3,4-dihydroxyphenyl glycol [DHPG], 5-hydroxyindoleacetic acid [5-HIAA], 3,4-dihydroxyphenylalanine [DOPA], and 3,4-dihydroxyphenylacetic acid [DOPAC]) in the CSF (CSF biomarkers) will be analyzed to evaluate the pharmacodynamic effect of JNJ-64140284.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Clinical Pharmacology Unit, Merksem, Belgium